CLINICAL TRIAL: NCT03864302
Title: Effect of Motor-imagery in Simulator-based Training in Transurethral Resection of Bladder Tumors - a Randomized Trial
Brief Title: Simulation in Transurethral Bladder Cancer Surgery
Acronym: OSATURB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Sarah Hjartbro Bube, Principal Investigator, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-19-1-OSATURB
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Virtual Reality; Education; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery (Experimental): The intervention group is informed about the concept of motor imagery (MI) for performance enhancement and are instructed in using the modified PETTLEP framework for TURB (table 1).(18) The intervention group performs a MI training session (MITS) prior to each VR simulation procedure.
  Table 1: PEELP framework:
  Physical: Sitting in front of the simulator, aloud to touch and move the scope Environment: Simulated sounds from the OR, including electrical device feedback from devices and vital measures Task: Four standardized TURB cases Timing: Each MI session is temporal to a simulated TURB case, max. 10 minutes Learning: Think aloud the major steps of the procedure using Emotions: Imagine the emotions when the surgery progresses and when an adverse event occurs Perspectives: Internal perspective thinking "then I…"
  Interventions: Behavioral: Motor Imagery
- Control (No Intervention): The control group proceeds directly to standard VR-simulator training.

INTERVENTIONS:
Behavioral: Motor Imagery — Motor imagery (MI) is a psychological technique for improvement of motor skills.(24) MI skill training (MIST) has been used and explored in several disciplines including Sports, Music, Education, Psychology and Medicine.(18) The literature has found positive effects on performances in professional athletes but also on rehabilitation of stroke patients.(25,26) MI is a cognitive imagery of a physical performance, e.g. a high jumper imagine a high jump, prior to performance. MI is not as effective as physical practice, but more effective compared to no training.(27) Further, MI combined with physical practice has been found to be more effective in skill performance in sports compared to physical practice alone.(18) MIST has shown promising results on surgical performances in flexible cystoscopy performed by doctors.(28)
  Arms: Motor Imagery

SUMMARY:
Bladder cancer (BC) is the seventh most common cancer disease among men worldwide, and the fourth most common cancer in Danish men with an incidence of more than 2000 and a prevalence of 650 per 100000 citizens.

BC have a poor prognosis even when treated radically with cystectomy. The 5-year survival rate after radical cystectomy for T2 muscle-invasive tumors are 23-60 % and decreasing further to 23 % for T4 muscle-invasive tumors. BC is highly recurrent with an overall recurrence of 50 %.

BC is considered to be the number one cost-expensive malignant disease of all malignant diseases measured by lifetime per patient in the United States.

The degree of muscle invasion in the bladder is histologically and clinically defined by a transurethral resection of the bladder tumor (TUR-B). The tumor is resected radically if possible.

Thus, it is of absolute importance that a sufficient TURB is performed, since a resection to the muscle layer of the bladder wall, the detrusor, is of prognostic value for the patient.

Problem: The quality of the surgery is depending on the surgeon A recent international meta-analysis shows that up to 78% of the tumors are not radically resected. When these tumors are resected in a second TURB 24-28% of the tumors are found to be muscle-invasive.

Furter, there is evidence indicating that the outcome of the resection is dependent on surgeon experience.

Large multi-centre retrospective studies have showed that resident-involvement in TURB results in less radical bladder tumor resections and result in higher recurrence rates of bladder tumors and high numbers of re-admission after TURB.

In Denmark, the current surgical curriculum states that TURB is a learning goal in the first year of the training. The formal training in TURB in Denmark is traditional apprenticeship in accordance with the Halstedian principle "see one, do one, teach one". No validated simulator-based certification in TURB exits today in Denmark or internationally.

Purpose: Start from the beginning - improve the training of the surgeons Simulator-based training in surgical procedures is an effective method to gain surgical skills in a large spectrum of surgical procedures. In the initial phase of the learning curve it has even proven more effective than traditional apprenticeship and thus both the World Health Organization (WHO) and the European Association of Urology (EAU) calls for implementation of simulation training programmes in medical surgical education.

The aim of this project is to validate and develop a simulator-based urological training programme in TURB, to implement the programme nationally and internationally, and hereby improve the outcomes in the surgical treatment of patients with bladder cancer.

DETAILED DESCRIPTION:
Doctors' surgical skills have consequences for patients outcomes and continued training and assessment of surgeons has the potential to improve patient safety and shorten learning curves in the operation room.

Traditionally, surgeons have acquired their skills by observation, supervision and direction of masters in the field. Such education is indispensable. Only, with the increasing demands on production, patient safety issues and decreasing working hours a need for alternatives to the classical surgical training has awoken.

Simulated surgeries make it possible to repeat and perfect performances until reaching a proficient level. Virtual reality (VR) simulators can provide continuously automated feedback while the doctor is performing the procedure and thus direct the training.

Thus, in the last decades simulators for surgical skills training have gained increasing popularity. Simulation training has been found efficient in skills acquisition in a variety of surgical procedures.Simulators allow repeating training until reaching a proficiency level in the skill. Ultimately, the doctor reaches a minimum competent skill acquisition in the procedure prior to advancing to surgeries on patients.

Mastery Learning (ML) is a strict proficiency training concept, in which the learner trains until reaching a minimum acquisition level. The endpoint of the training is hereby a predefined competency level, and not an arbitrary amount of training hours. Hence, ML ensures a minimum skill acquisition level.

In the initial learning phase of the learning curve the use of ML simulation training has been proven superior to traditional apprenticeship.

To identify proficiency, assessments are needed. The assessments should be based on solid evidence of validity. The development and validation of tests are essential in a proficiency-based curriculum.

Constructing a training curriculum in surgery should be based on a defined framework. Zevin et al. proposed a training-design framework composed of three steps: cognitive knowledge (conceptualization, visualization and verbalization), psychomotor skills training (deliberate and distributed self-regulated training to a targeted proficiency-level, with continuing feedback and maintenance) and non-technical skills (communication, collaboration, professionalism and management). Thomas et al. proposed a six-step approach for curriculum development including problem identification, need assessment, goal setting and teaching objectives, educational strategies, implementation and evaluation and feedback.

A needs assessment analysis among residents and urologists in Denmark from 2017 confirms the feasibility and necessity of comprehensive ex-vivo simulation-based curriculum in TUR-B. TUR-B simulators have been available for a decade but some have proven insufficiency, others promising, but there is a need for creation of evidence-based simulator training programs and development of valid assessments tool to evaluate the performances.

The effect on training of a novel curriculum can be explored and evaluated using a framework such as Kirkpatrick's model for evaluation of training effect on skills, transfer from simulation to workplace, benefits for patients, and finally economics and return of investments.

This trial aims to develop an evidence-based TURB training and certification program including an assessment tool for clinical procedures (trial 1.1), learning curve study (trial 1.2) and pre- and post-training study and effects on operation room TURB performance (trial 1.3) and explore the prognostic clinical value of performance on simulation-based test (trial 1.4).

ELIGIBILITY:
Inclusion Criteria:

* Doctors
* Informed written consent.
* Four video-recordings of TURBs.

Exclusion Criteria:

* Not providing four video recordings of TURB procedures
* Simulation-based training course in TURB within 6 months
* No consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
OSATURB total score | 8 hours pr. participant
  Assessment tool with nine items, each item i rated on a 5-point Likert scale, minimum of 1, max. 5.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bube, MD, Principal Investigator — Zeland Region
Locations (1):
- Urology Department Zealand University Hospital, Roskilde, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birkmeyer JD, Finks JF, O'Reilly A, Oerline M, Carlin AM, Nunn AR, Dimick J, Banerjee M, Birkmeyer NJ; Michigan Bariatric Surgery Collaborative. Surgical skill and complication rates after bariatric surgery. N Engl J Med. 2013 Oct 10;369(15):1434-42. doi: 10.1056/NEJMsa1300625. PMID 24106936
- [Background] Bjerrum F, Thomsen ASS, Nayahangan LJ, Konge L. Surgical simulation: Current practices and future perspectives for technical skills training. Med Teach. 2018 Jul;40(7):668-675. doi: 10.1080/0142159X.2018.1472754. Epub 2018 Jun 17. PMID 29911477
- [Background] Cook DA, Hatala R, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hamstra SJ. Technology-enhanced simulation for health professions education: a systematic review and meta-analysis. JAMA. 2011 Sep 7;306(9):978-88. doi: 10.1001/jama.2011.1234. PMID 21900138
- [Background] McGaghie WC, Issenberg SB, Barsuk JH, Wayne DB. A critical review of simulation-based mastery learning with translational outcomes. Med Educ. 2014 Apr;48(4):375-85. doi: 10.1111/medu.12391. PMID 24606621
- [Background] McGaghie WC, Issenberg SB, Cohen ER, Barsuk JH, Wayne DB. Does simulation-based medical education with deliberate practice yield better results than traditional clinical education? A meta-analytic comparative review of the evidence. Acad Med. 2011 Jun;86(6):706-11. doi: 10.1097/ACM.0b013e318217e119. PMID 21512370
- [Background] Konge L, Clementsen PF, Ringsted C, Minddal V, Larsen KR, Annema JT. Simulator training for endobronchial ultrasound: a randomised controlled trial. Eur Respir J. 2015 Oct;46(4):1140-9. doi: 10.1183/13993003.02352-2015. Epub 2015 Jul 9. PMID 26160875
- [Background] Borgersen NJ, Naur TMH, Sorensen SMD, Bjerrum F, Konge L, Subhi Y, Thomsen ASS. Gathering Validity Evidence for Surgical Simulation: A Systematic Review. Ann Surg. 2018 Jun;267(6):1063-1068. doi: 10.1097/SLA.0000000000002652. PMID 29303808
- [Background] Zevin B, Levy JS, Satava RM, Grantcharov TP. A consensus-based framework for design, validation, and implementation of simulation-based training curricula in surgery. J Am Coll Surg. 2012 Oct;215(4):580-586.e3. doi: 10.1016/j.jamcollsurg.2012.05.035. Epub 2012 Jul 3. PMID 22762990
- [Background] Nayahangan LJ, Bolling Hansen R, Gilboe Lindorff-Larsen K, Paltved C, Nielsen BU, Konge L. Identifying content for simulation-based curricula in urology: a national needs assessment. Scand J Urol. 2017 Dec;51(6):484-490. doi: 10.1080/21681805.2017.1352618. Epub 2017 Jul 26. PMID 28743217
- [Background] Schout BM, Bemelmans BL, Martens EJ, Scherpbier AJ, Hendrikx AJ. How useful and realistic is the uro trainer for training transurethral prostate and bladder tumor resection procedures? J Urol. 2009 Mar;181(3):1297-303; discussion 1303. doi: 10.1016/j.juro.2008.10.169. Epub 2009 Jan 18. PMID 19152928
- [Background] de Vries AH, van Genugten HG, Hendrikx AJ, Koldewijn EL, Schout BM, Tjiam IM, van Merrienboer JJ, Muijtjens AM, Wagner C. The Simbla TURBT Simulator in Urological Residency Training: From Needs Analysis to Validation. J Endourol. 2016 May;30(5):580-7. doi: 10.1089/end.2015.0723. Epub 2016 Jan 22. PMID 26671712
- [Background] Cook DA. Twelve tips for evaluating educational programs. Med Teach. 2010;32(4):296-301. doi: 10.3109/01421590903480121. PMID 20353325
- [Background] Feldman M, Lazzara EH, Vanderbilt AA, DiazGranados D. Rater training to support high-stakes simulation-based assessments. J Contin Educ Health Prof. 2012 Fall;32(4):279-86. doi: 10.1002/chp.21156. PMID 23280532
- [Background] Downing SM, Haladyna TM. Validity threats: overcoming interference with proposed interpretations of assessment data. Med Educ. 2004 Mar;38(3):327-33. doi: 10.1046/j.1365-2923.2004.01777.x. PMID 14996342
- [Background] Feltz DL, Landers DM. The Effects of Mental Practice on Motor Skill Learning and Performance: A Meta-analysis. J Sport Psychol. 1983 Mar;5(1):25-57.
- [Background] Schuster C, Hilfiker R, Amft O, Scheidhauer A, Andrews B, Butler J, Kischka U, Ettlin T. Best practice for motor imagery: a systematic literature review on motor imagery training elements in five different disciplines. BMC Med. 2011 Jun 17;9:75. doi: 10.1186/1741-7015-9-75. PMID 21682867
- [Background] Rasmussen KMB, Hertz P, Laursen CB, Arshad A, Saghir Z, Clementsen PF, Konge L. Ensuring Basic Competence in Thoracentesis. Respiration. 2019;97(5):463-471. doi: 10.1159/000495686. Epub 2019 Jan 9. PMID 30625480
- [Background] Cook DA, Hamstra SJ, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hatala R. Comparative effectiveness of instructional design features in simulation-based education: systematic review and meta-analysis. Med Teach. 2013;35(1):e867-98. doi: 10.3109/0142159X.2012.714886. Epub 2012 Sep 3. PMID 22938677
- [Background] McGaghie WC, Miller GE, Sajid AW, Telder TV. Competency-based curriculum development on medical education: an introduction. Public Health Pap. 1978;(68):11-91. No abstract available. PMID 664734
- [Background] Cook DA, Zendejas B, Hamstra SJ, Hatala R, Brydges R. What counts as validity evidence? Examples and prevalence in a systematic review of simulation-based assessment. Adv Health Sci Educ Theory Pract. 2014 May;19(2):233-50. doi: 10.1007/s10459-013-9458-4. Epub 2013 May 2. PMID 23636643
- [Background] Thomas MR, Beckman TJ, Mauck KF, Cha SS, Thomas KG. Group assessments of resident physicians improve reliability and decrease halo error. J Gen Intern Med. 2011 Jul;26(7):759-64. doi: 10.1007/s11606-011-1670-4. Epub 2011 Mar 3. PMID 21369769
- [Background] Holmes PS, Collins DJ. The PETTLEP Approach to Motor Imagery: A Functional Equivalence Model for Sport Psychologists. J Appl Sport Psyholgy. 2001;13(1):60-83.
- [Background] Olsson CJ, Jonsson B, Larsson A, Nyberg L. Motor representations and practice affect brain systems underlying imagery: an FMRI study of internal imagery in novices and active high jumpers. Open Neuroimag J. 2008;2:5-13. doi: 10.2174/1874440000802010005. Epub 2008 Jan 31. PMID 19018312
- [Background] Riccio I, Iolascon G, Barillari MR, Gimigliano R, Gimigliano F. Mental practice is effective in upper limb recovery after stroke: a randomized single-blind cross-over study. Eur J Phys Rehabil Med. 2010 Mar;46(1):19-25. PMID 20332722
- [Background] Komesu Y, Urwitz-Lane R, Ozel B, Lukban J, Kahn M, Muir T, Fenner D, Rogers R. Does mental imagery prior to cystoscopy make a difference? A randomized controlled trial. Am J Obstet Gynecol. 2009 Aug;201(2):218.e1-9. doi: 10.1016/j.ajog.2009.04.008. Epub 2009 May 30. PMID 19481728
- [Background] Ostergaard ML, Rue Nielsen K, Albrecht-Beste E, Kjaer Ersboll A, Konge L, Bachmann Nielsen M. Simulator training improves ultrasound scanning performance on patients: a randomized controlled trial. Eur Radiol. 2019 Jun;29(6):3210-3218. doi: 10.1007/s00330-018-5923-z. Epub 2019 Jan 7. PMID 30617476
- [Background] Knol MJ, Pestman WR, Grobbee DE. The (mis)use of overlap of confidence intervals to assess effect modification. Eur J Epidemiol. 2011 Apr;26(4):253-4. doi: 10.1007/s10654-011-9563-8. Epub 2011 Mar 19. No abstract available. PMID 21424218
- [Background] Dunn W, Dong Y, Zendejas B, Ruparel R, Farley D. Simulation, Mastery Learning and Healthcare. Am J Med Sci. 2017 Feb;353(2):158-165. doi: 10.1016/j.amjms.2016.12.012. Epub 2016 Dec 16. PMID 28183417
- [Background] Ericsson KA. Acquisition and maintenance of medical expertise: a perspective from the expert-performance approach with deliberate practice. Acad Med. 2015 Nov;90(11):1471-86. doi: 10.1097/ACM.0000000000000939. PMID 26375267
- [Background] Woehr DJ, Huffcutt AI. Rater training for performance appraisal: A quantitative review. J Occup Organ Psychol. 1994 Sep;67(3):189-205.
- [Derived] Bube SH, Kingo PS, Madsen MG, Vasquez JL, Norus T, Olsen RG, Dahl C, Hansen RB, Konge L, Azawi N. National Implementation of Simulator Training Improves Transurethral Resection of Bladder Tumours in Patients. Eur Urol Open Sci. 2022 Apr 1;39:29-35. doi: 10.1016/j.euros.2022.03.003. eCollection 2022 May. PMID 35528788
- [Derived] Bube SH, Kingo PS, Madsen MG, Vasquez JL, Norus T, Olsen RG, Dahl C, Hansen RB, Konge L, Azawi N. Validation of a Novel Assessment Tool Identifying Proficiency in Transurethral Bladder Tumor Resection: The OSATURBS Assessment Tool. J Endourol. 2022 Apr;36(4):572-579. doi: 10.1089/end.2021.0768. PMID 34731011